CLINICAL TRIAL: NCT05592730
Title: Antimullerian Hormone Receptor 2 Polymorphism in Blood and Granulosa Cells in Unexplained Infertility
Brief Title: AMHR2 Polymorphism in Blood and Granulosa Cells in Unexplained Infertility
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.06.2022-E.65396
Record Dates: First submitted 2022-10-20; First posted 2022-10-25 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Infertility, Female; AMH; IVF
Keywords: unexplained infertility; anti-mullerian hormone receptor2 polymorphism
MeSH Terms: conditions — Infertility, Female | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Study Group: Patients with Unexplained İnfertility
  Interventions: Genetic: AMHR2 polymorphism in blood; Genetic: AMHR2 polymorphism in granulosa cell
- First Control Group: Healthy Multiparous Women
  Interventions: Genetic: AMHR2 polymorphism in blood
- Second Control Group: A: Patients with male infertility B: Patients with tubal factor
  Interventions: Genetic: AMHR2 polymorphism in blood; Genetic: AMHR2 polymorphism in granulosa cell

INTERVENTIONS:
Genetic: AMHR2 polymorphism in blood — 1 tube of blood taken at the first application
Genetic: AMHR2 polymorphism in granulosa cell — Extraction of granulosa cell from the follicle fluid obtained during OPU
  Groups: Second Control Group; Study Group

SUMMARY:
There are various known parameters for assessing ovarian reserve, including ovarian volume, antral follicle count, follicle stimulating hormone (FSH) and Inhibin B at the beginning of the menstrual cycle, as well as anti-Mullerian hormone (AMH). Anti-müllerian hormone is a dimeric glycoprotein and a member of the transforming growth factor β family that plays a role in the regulation of follicular development. AMH is produced by granulosa cells of the early developing follicles in the ovary, and continues to be expressed in the growing follicles until these follicles have reached a size of 4-6 mm and a differentiation state at which AMH becomes receptive for exogenous FSH, and may be selected for dominance.It exerts its biological effects through the receptor AMHR2, which is present on granulosa and theca cells. Considering the important role of the AMH signalling pathway in regulating FSH sensitivity in the ovary and follicular recruitment and selection, it is appropriate to consider that variation in the genes encoding key proteins in the pathway may influence ovarian response. The aim of this study is to investigate the effect of the distribution of single gene polymorphisms of the AMHR2 receptor gene A-482G/rs200255 in patients with unexplained infertility and to compare this distribution with the distribution in women without infertility.

DETAILED DESCRIPTION:
This prospective, controlled cohort study was conducted at IVF Centre of Department of Obstetrics and Gynecology, Bezmialem University Hospital between October 2022 and April 2023. The study protocol was approved by the Ethical Committee of the Medical Faculty of Bezmialem University. Written informed consent was obtained from all patients. This trial was designed and reported according to the Consolidated Standards of Reporting Trials (CONSORT) guidelines.

The patients were divided into 3 groups. Group 1 (study group; unexplained infertilitiy, n=32), Group 2 ( first control group; healthy women with a history of at least one successful previous pregnancy, n=32), Group 3 ( second control group; infertile patients undergo IVF because of male or tubal factor, n=32). Inclusion criteria for the study were as follows: <40 years of age, normal serum levels of TSH and prolactin presence of both ovaries without any morphological abnormalities, normal ovulatory cycles (25-35 days), body mass index (BMI) ≤30, no previous history of poor response and no evidence of endocrine disease, such as polycystic ovary syndrome, hipo-hyper prolactinemia, no use of hormone therapy in the 6 months preceding the recruitment and commencing IVF treatment. Patients with moderate/severe endometriosis (stage III and IV), previous ovarian surgery or underwent chemo/radiotherapy excluded from the study.

At the first application, peripheral blood will be taken from the Study group, 1st Control and 2nd Control group to evaluate polymorphisms of the AMHR2-482A>G(rs200255) with PCR analysis. During IVF treatment at the day of ovum pick up; follicular fluid will be collected to isolate granulosa cell for polymorphisms of the AMHR2-482A>G(rs200255) with PCR analysis.

The total number of embryos, the number of embryos transferred, the number of frozen and viable embryos will be recorded. After the embryo transfer is performed in the study group and the 2nd control group, the pregnancy results will be recorded by checking the bhcg in the blood on the 10-12th day of the transfer.

ELIGIBILITY:
inclusion criteria

* unexplained infertility (study group)
* a healthy women with a history of at least one successful previous pregnancy resulting from spontaneous conception (first control group)
* infertility caused by male factor, tubal factor (second control group)
* <40 years of age
* normal serum levels of TSH and prolactin
* presence of both ovaries without any morphological abnormalities
* normal ovulatory cycles (25-35 days)
* body mass index (BMI) ≤30
* no previous history of poor response and no evidence of endocrine disease, such as polycystic ovary syndrome, hipo-hyper prolactinemia
* no use of hormone therapy in the 6 months preceding the recruitment
* undergoing IVF

exclusion criteria

* Patients with moderate/severe endometriosis (stage III and IV)
* previous ovarian surgery or underwent chemo/radiotherapy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Unexplained infertility group
Sampling Method: Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Ovarian response | average of 6 months
  Number of oocytes, 5th day blast rate

SECONDARY OUTCOMES:
Ongoing pregnancy rate | average of 9 months
  Pregnancies that continue until the 12th week of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Pinar Ozcan, MD, PhD, Study Chair — BEZMİALEM VAKIF ÜNİVERSİTESİ
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yoshida Y, Yamashita Y, Saito N, Ono Y, Yamamoto H, Nakamura Y, Hayashi A, Terai Y, Ohmichi M. Analyzing the possible involvement of anti-Mullerian hormone and anti-Mullerian hormone receptor II single nucleotide polymorphism in infertility. J Assist Reprod Genet. 2014 Feb;31(2):163-8. doi: 10.1007/s10815-013-0134-7. Epub 2013 Nov 24. PMID 24271023
- [Background] Peluso C, Fonseca FL, Gastaldo GG, Christofolini DM, Cordts EB, Barbosa CP, Bianco B. AMH and AMHR2 polymorphisms and AMH serum level can predict assisted reproduction outcomes: a cross-sectional study. Cell Physiol Biochem. 2015;35(4):1401-12. doi: 10.1159/000373961. Epub 2015 Mar 12. PMID 25790842
- [Background] Cerra C, Newman WG, Tohlob D, Byers H, Horne G, Roberts SA, Mohiyiddeen L. AMH type II receptor and AMH gene polymorphisms are not associated with ovarian reserve, response, or outcomes in ovarian stimulation. J Assist Reprod Genet. 2016 Aug;33(8):1085-91. doi: 10.1007/s10815-016-0711-7. Epub 2016 May 3. PMID 27142041